CLINICAL TRIAL: NCT01715532
Title: Phase II Study of Huachansu for Treatment of Advanced Hepatocellular Carcinoma and the Correlation With Na+/K+-ATPase
Brief Title: Role of Huachansu in Treating Hepatocellular Carcinoma and the Correlation With Na+/K+-ATPase
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hao Chen, Associated Professor, MD, Ph D, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCS-2012
Record Dates: First submitted 2012-08-17; First posted 2012-10-29 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Huachansu; Na+/K+-ATPase α3; transcatheter arterial chemoembolization; randomized controlled trial
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — huachansu

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huachansu + TACE (Experimental): Patients in this arm will receive Huachansu tablets each 3 and 3 times a day orally, as well as transcatheter arterial chemoembolization every 4 weeks, until progression of disease or adverse effects leading to termination of treatment. Each 4-week period is one cycle of treatment.
  Interventions: Drug: Huachansu; Other: TACE
- TACE (Active Comparator): Patients in this arm will receive transcatheter arterial chemoembolization every 4 weeks, until progression of disease or adverse effects leading to termination of treatment. Each 4-week period is one cycle of treatment.
  Interventions: Other: TACE

INTERVENTIONS:
Drug: Huachansu
  Arms: Huachansu + TACE
Other: TACE
  Other Names: transcatheter arterial chemoembolization

SUMMARY:
Primary Outcome Measures:

- To compare the progression free survival(PFS) in patients with unresectable hepatocellular carcinoma(HCC) treated with transcatheter arterial chemoembolization(TACE) with or without Huachansu, and the correlation between PFS and expression of peripheral Na+/K+-ATPase α3 family.

Secondary Outcome Measures:

- To compare the overall survival(OS), objective response rate(ORR), and side effects of treating HCC with TACE plus Huachansu or TACE alone.

Exploratory Outcome Measures:

- To evaluate the correlation between prognosis and expression of peripheral Na+/K+-ATPase α3 family.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-75 years of age.
* Diagnosis of hepatocellular carcinoma. Biopsy is the preferred method of diagnosis (option 1). As far as clinically possible, the results of a biopsy should be obtained to confirm the diagnosis prior to the initiation of investigational product administration.. Non-biopsy criteria are allowed in cases where a biopsy result is unavailable and a biopsy procedure is not clinically indicated (option 2). (Option 1: Biopsy-proven HCC (histology or cytology); Option 2 - patient must fulfill the following criteria: i. Radiological evidence of HCC showing lesion arterial hypervascularity and venous phase washout by either dynamic (triple-phase), contrast-enhanced computed tomography of the abdomen OR dynamic (triple-phase) contrast (gadolinium)-enhanced MRI, AND ii. Serology positive for hepatitis B or C, AND iii. Alpha fetoprotein > 400 μg/L at the time of diagnosis.)
* No metastasis outside liver.
* Unable or unwilling to receive radical surgery.
* No prior transcatheter arterial chemoembolization.
* No prior treatment of bufalins including Huachansu.
* At least one measurable untreated lesion. All subjects must have at least one measurable lesion unidimensionally by CT or MRI scan, according to modified RECIST for HCC, that has not been previously treated with surgery, irradiation, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* Cirrhotic status of Child-Pugh Class A or B.
* Adequate hematologic function with absolute neutrophil counts ≥ 1.5×109 /L, platelet count ≥ 50 x 109/L, and hemoglobin ≥ 85 g/L.
* Signed Written Informed Consent.
* Subjects who have a life expectancy of at least 3 months.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study that the risk of pregnancy is minimized.

Exclusion Criteria:

* Previously treated target lesion with irradiation, TACE, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* Cirrhotic status of Child-Pugh Class C.
* Severe diseases of heart, liver, kidney, etc that may cause inadequate organ functions
* History of other malignant tumor in 5 years.
* Pregnant or lactating women.
* Mentally disordered.
* Participation of other clinical trials within a month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, MD, Ph D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao H, He J, Cheng CS, Zhuang L, Chen H, Meng Z. Unresectable hepatocellular carcinoma: transarterial chemoembolisation plus Huachansu - a single-center randomised controlled trial. BMJ Support Palliat Care. 2023 Jul 3;14(e2):e003870. doi: 10.1136/spcare-2022-003870. Online ahead of print. PMID 37400162